CLINICAL TRIAL: NCT07271472
Title: Total Intravenous Anesthesia (TIVA), Combined Intravenous-Volatile Anesthesia (CIVA), and Balanced Anesthesia (BAL) on Perioperative Oxidative Stress in Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: Oxidative Stress Effects of TIVA, CIVA, and Balanced Anesthesia in VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Oral Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATAUNIVATS
Record Dates: First submitted 2025-11-25; First posted 2025-12-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: VATS; Video Assisted Thoracoscopic Surgery
Keywords: Video-Assisted Thoracoscopic Surgery; Total Intravenous Anesthesia; Combined Intravenous Volatile Anesthesia; Balanced Anesthesia; Malondialdehyde; Total Oxidant Status; Total Antioxidant Status; Superoxide Dismutase
MeSH Terms: interventions — Population Groups; Balanced Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total Intravenous Anesthesia (TIVA) Group (Experimental): Anesthesia induction will include 2 mg midazolam, 2-2.5 mg/kg propofol, 0.6-0.9 mg/kg rocuronium, and 1 μg/kg remifentanil. Maintenance will be provided with target-controlled infusion (TCI) propofol at a Ce of 4-6 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL while maintaining the bispectral index (BIS) between 40-60.
  Interventions: Drug: Total Intravenous Anesthesia (TIVA) Group
- Balanced Anesthesia (BAL) Group (Experimental): Induction will follow the same protocol as the TIVA group. During maintenance, desflurane 5-7% (MAC 1-1.3) and TCI remifentanil at a Ce of 1.5-3 ng/mL will be administered, targeting a BIS value between 40-60.
  Interventions: Drug: Balanced Anesthesia (BAL) Group
- Combined Intravenous Volatile Anesthesia (CIVA) Group (Experimental): Induction will follow the same protocol as other groups. Maintenance will include TCI propofol at a Ce of 2-4 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL along with 3% desflurane (MAC 0.5), keeping BIS values between 40-60.
  Interventions: Drug: Combined Intravenous Volatile Anesthesia

INTERVENTIONS:
Drug: Total Intravenous Anesthesia (TIVA) Group — Anesthesia induction will include 2 mg midazolam, 2-2.5 mg/kg propofol, 0.6-0.9 mg/kg rocuronium, and 1 μg/kg remifentanil. Maintenance will be provided with target-controlled infusion (TCI) propofol at a Ce of 4-6 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL while maintaining the bispectral index (BIS) between 40-60.
  Other Names: TIVA Group
  Arms: Total Intravenous Anesthesia (TIVA) Group
Drug: Balanced Anesthesia (BAL) Group — Induction will follow the same protocol as the TIVA group. During maintenance, desflurane 5-7% (MAC 1-1.3) and TCI remifentanil at a Ce of 1.5-3 ng/mL will be administered, targeting a BIS value between 40-60.
  Other Names: BAL Group
  Arms: Balanced Anesthesia (BAL) Group
Drug: Combined Intravenous Volatile Anesthesia — Induction will follow the same protocol as other groups. Maintenance will include TCI propofol at a Ce of 2-4 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL along with 3% desflurane (MAC 0.5), keeping BIS values between 40-60.
  Other Names: CIVA Group
  Arms: Combined Intravenous Volatile Anesthesia (CIVA) Group

SUMMARY:
The primary objective of our study is to compare the effects of total intravenous anesthesia (TIVA), combined intravenous-volatile anesthesia (CIVA), and balanced anesthesia (BAL) methods on perioperative oxidative stress parameters, such as Malondialdehyde (MDA), Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and Superoxide Dismutase (SOD), in patients undergoing video-assisted thoracoscopic surgery (VATS). The secondary objective is to record perioperative vital parameters, arterial blood gas values obtained at specific stages of the surgery, and the incidence of postoperative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
Scientific Rationale and Validity of the Medical Research Hypoxic pulmonary vasoconstriction (HPV) is a homeostatic mechanism unique to the pulmonary vascular system. In response to alveolar hypoxia, intrapulmonary arteries constrict and redirect blood flow toward better-oxygenated lung segments, thereby optimizing ventilation/perfusion matching and systemic oxygenation . Additionally, HPV acts as a physiological protective mechanism by reducing the shunt of deoxygenated blood and improving the degree of hypoxemia. This physiological modulation is influenced by various factors including medications, temperature, acid-base status, airway pressure, patient positioning, and cardiac output . Numerous animal and isolated lung studies have demonstrated that HPV is modulated by volatile anesthetics . However, human studies have reported inconsistent results regarding the effects of various anesthetics on systemic oxygenation during one-lung ventilation.

One-lung ventilation is frequently employed during thoracic surgical procedures such as thoracotomy and thoracoscopy to provide an adequate surgical view. Patients undergoing one-lung ventilation are at risk of hypoxemia due to impaired oxygenation, as well as postoperative lung injury attributable to oxidative damage occurring during reventilation of the non-dependent lung.

During one-lung ventilation, the non-ventilated lung becomes not only atelectatic but also hypoperfused as a result of HPV. Once two-lung ventilation is re-established, the reintroduction of oxygen into the airways triggers reactive pulmonary vasodilation and reperfusion of the lung tissue, which may result in the generation of excessive oxidative radicals. Although the lung is relatively resistant to hypoxia owing to dual blood supply and consumption of oxygen stored in alveolar spaces, re-expansion injury observed after pneumothorax treatment and reperfusion injury following lung transplantation serve as examples of potential oxidative damage .

Research Questions How do TIVA, CIVA, and BAL anesthetic techniques affect oxidative stress responses in patients undergoing one-lung ventilation? Which anesthetic management approach (CIVA, TIVA, BAL) provides better preservation of oxygenation? Will there be a significant difference in postoperative nausea and vomiting (PONV) incidence among the groups? Study Design, Methods, and Procedures Participants Written informed consent will be obtained from all participants. Sixty patients aged 18-65 years, classified as American Society of Anesthesiologists (ASA) Physical Status I-II, scheduled for elective video-assisted thoracoscopic surgery (VATS) at Atatürk University Medical Faculty Hospital between December 1, 2025 and May 1, 2026, and requiring one-lung ventilation for more than 60 minutes will be included. Patients will be informed about the study prior to enrollment. Individuals who decline participation, have known allergies to the study drugs, have a recent history of vitamin supplementation, or who have significant cardiovascular, renal, or hepatic disease will be excluded. The study will be conducted in three groups.

Randomization Patients will be randomly assigned into three equal groups (TIVA, CIVA, and BAL) using the Microsoft Excel RAND function. All other investigators and outcome assessors will remain blinded to group allocation.

Total Intravenous Anesthesia (TIVA) Group Anesthesia induction will include 2 mg midazolam, 2-2.5 mg/kg propofol, 0.6-0.9 mg/kg rocuronium, and 1 μg/kg remifentanil. Maintenance will be provided with target-controlled infusion (TCI) propofol at a Ce of 4-6 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL while maintaining the bispectral index (BIS) between 40-60.

Balanced Anesthesia (BAL) Group Induction will follow the same protocol as the TIVA group. During maintenance, desflurane 5-7% (MAC 1-1.3) and TCI remifentanil at a Ce of 1.5-3 ng/mL will be administered, targeting a BIS value between 40-60.

Combined Intravenous-Volatile Anesthesia (CIVA) Group Induction will follow the same protocol as other groups. Maintenance will include TCI propofol at a Ce of 2-4 μg/mL and TCI remifentanil at a Ce of 1.5-3 ng/mL along with 3% desflurane (MAC 0.5), keeping BIS values between 40-60.

Perioperative Monitoring and Sample Collection Upon arrival to the operating room, standard monitoring (ECG and SpO₂) will be applied. A 20G radial arterial catheter will be inserted under sterile conditions for continuous invasive blood pressure monitoring and blood sampling.

Following induction, patients will be intubated using an appropriately sized (35Fr, 37Fr, or 39Fr) Robertshaw double-lumen endotracheal tube. Position verification will be conducted with a fiberoptic bronchoscope before and after lateral positioning. Pressure-controlled volume-guaranteed (PCV-VG) ventilation will be used during both two-lung and one-lung ventilation with PEEP set at 5 cmH₂O. During one-lung ventilation, tidal volume will be set at 4-6 mL/kg keeping peak inspiratory pressure <30 cmH₂O, FiO₂ between 0.6-1.0 to maintain SpO₂ >90%, and respiratory rate adjusted to ensure normocapnia.

Blood samples for measurement of oxidative stress markers-Malondialdehyde (MDA), Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and Superoxide Dismutase (SOD)-will be drawn from the arterial catheter at three time points:

T1: Before anesthesia induction T2: Before re-establishing two-lung ventilation T3: 30 minutes after re-establishing two-lung ventilation Samples will be centrifuged at +4°C, 4500 rpm for 7 minutes. The obtained serum will be stored at -80°C in Eppendorf tubes until analysis. Serum levels will be determined using the ELISA method. Recorded values will be transferred to Excel spreadsheets for evaluation and statistical processing.

During anesthesia, at 15, 30, 45, and 60 minutes of one-lung ventilation and 30 minutes after resuming two-lung ventilation, TCI remifentanil dose, TCI propofol dose, minimum alveolar concentration (MAC), peak inspiratory pressure (Ppeak), BIS values, heart rate, and mean arterial pressure will be recorded. Arterial blood gas samples will be routinely obtained. After extubation, patients will be transferred to the post-anesthesia care unit (PACU) and evaluated for postoperative nausea and vomiting (PONV) at the 30th minute.

Statistical Analysis Statistical analyses will be performed using SPSS Statistics Version 22 (IBM, Armonk, NY, USA). Normality will be assessed with the Kolmogorov-Smirnov test. Normally distributed variables will be analyzed using the Student's t-test, whereas non-normally distributed variables will be evaluated using the Mann-Whitney U test. A p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years,
* American Society of Anesthesiologists (ASA) Physical Status Class I-II,
* Scheduled for elective Video-Assisted Thoracoscopic Surgery (VATS)
* Requiring one-lung ventilation for more than 60 minutes

Exclusion Criteria:

* Refusal to participate in the study
* History of allergy to the drugs to be used
* Recent history of vitamin supplementation
* History of severe cardiac, renal, or hepatic disease
* ASA III-IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Malondialdehyde levels in perioperatively collected blood samples | Immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation
  For measurement of this marker, arterial blood samples will be collected from the radial artery at three time points: immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation. The collected blood samples will be centrifuged at +4 °C at 4500 rpm for 7 minutes. The obtained serum samples will be transferred into Eppendorf tubes and stored at -80 °C until the day of analysis. Serum levels of MDA will be measured using the ELISA method.
Total Antioxidant Status levels in perioperatively collected blood samples | Immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation
  For measurement of this marker, arterial blood samples will be collected from the radial artery at three time points: immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation. The collected blood samples will be centrifuged at +4 °C at 4500 rpm for 7 minutes. The obtained serum samples will be transferred into Eppendorf tubes and stored at -80 °C until the day of analysis. Serum levels of TAS will be measured using the ELISA method.
Total Oxidant Status levels in perioperatively collected blood samples | Immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation
  For measurement of this marker, arterial blood samples will be collected from the radial artery at three time points: immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation. The collected blood samples will be centrifuged at +4 °C at 4500 rpm for 7 minutes. The obtained serum samples will be transferred into Eppendorf tubes and stored at -80 °C until the day of analysis. Serum levels of TOS will be measured using the ELISA method.
Superoxide Dismutase levels in perioperatively collected blood samples | Immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation
  For measurement of this marker, arterial blood samples will be collected from the radial artery at three time points: immediately before anesthesia induction, before the transition from one-lung ventilation to two-lung ventilation, and 30 minutes after the re-establishment of two-lung ventilation. The collected blood samples will be centrifuged at +4 °C at 4500 rpm for 7 minutes. The obtained serum samples will be transferred into Eppendorf tubes and stored at -80 °C until the day of analysis. Serum levels of SOD will be measured using the ELISA method.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | From 1 to 24 hour post operatively
  Incidence of post operative nausea and vomiting (PONV)
Partial pressure of oxygen (PaO₂) values | During anesthesia induction, at 15, 30, 45, and 60 minutes of one-lung ventilation, and 30 minutes after the transition to two-lung ventilation
  Arterial blood gas samples will be obtained during anesthesia induction, at 15, 30, 45, and 60 minutes of one-lung ventilation, and 30 minutes after the transition to two-lung ventilation, and the partial pressure of oxygen (PaO₂) values will be recorded.
Partial pressure of carbon dioxide pressure (PaCO₂) | During anesthesia induction, at 15, 30, 45, and 60 minutes of one-lung ventilation, and 30 minutes after the transition to two-lung ventilation
  Arterial blood gas samples will be obtained during anesthesia induction, at 15, 30, 45, and 60 minutes of one-lung ventilation, and 30 minutes after the transition to two-lung ventilation, and partial carbon dioxide pressure (PaCO₂) values will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Oral Ahiskalioglu, Professor, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy concerns and institutional regulations. Data will be securely stored and used solely for the purposes of this study and related scientific publications.

REFERENCES:
- [Result] Comhair SA, Erzurum SC. Antioxidant responses to oxidant-mediated lung diseases. Am J Physiol Lung Cell Mol Physiol. 2002 Aug;283(2):L246-55. doi: 10.1152/ajplung.00491.2001. PMID 12114185
- [Result] Lang JD, McArdle PJ, O'Reilly PJ, Matalon S. Oxidant-antioxidant balance in acute lung injury. Chest. 2002 Dec;122(6 Suppl):314S-320S. doi: 10.1378/chest.122.6_suppl.314s. PMID 12475808
- [Result] Cheng YJ, Chan KC, Chien CT, Sun WZ, Lin CJ. Oxidative stress during 1-lung ventilation. J Thorac Cardiovasc Surg. 2006 Sep;132(3):513-8. doi: 10.1016/j.jtcvs.2006.03.060. PMID 16935103
- [Result] Sharifian Attar A, Tabari M, Rahnamazadeh M, Salehi M. A comparison of effects of propofol and isoflurane on arterial oxygenation pressure, mean arterial pressure and heart rate variations following one-lung ventilation in thoracic surgeries. Iran Red Crescent Med J. 2014 Feb;16(2):e15809. doi: 10.5812/ircmj.15809. Epub 2014 Feb 8. PMID 24719749
- [Result] Xu WY, Wang N, Xu HT, Yuan HB, Sun HJ, Dun CL, Zhou SQ, Zou Z, Shi XY. Effects of sevoflurane and propofol on right ventricular function and pulmonary circulation in patients undergone esophagectomy. Int J Clin Exp Pathol. 2013 Dec 15;7(1):272-9. eCollection 2014. PMID 24427348
- [Result] Schwarzkopf K, Schreiber T, Preussler NP, Gaser E, Huter L, Bauer R, Schubert H, Karzai W. Lung perfusion, shunt fraction, and oxygenation during one-lung ventilation in pigs: the effects of desflurane, isoflurane, and propofol. J Cardiothorac Vasc Anesth. 2003 Feb;17(1):73-5. doi: 10.1053/jcan.2003.13. PMID 12635064
- [Result] Loer SA, Scheeren TW, Tarnow J. Desflurane inhibits hypoxic pulmonary vasoconstriction in isolated rabbit lungs. Anesthesiology. 1995 Sep;83(3):552-6. doi: 10.1097/00000542-199509000-00014. PMID 7661356
- [Result] Karzai W, Haberstroh J, Priebe HJ. Effects of desflurane and propofol on arterial oxygenation during one-lung ventilation in the pig. Acta Anaesthesiol Scand. 1998 Jul;42(6):648-52. doi: 10.1111/j.1399-6576.1998.tb05296.x. PMID 9689269
- [Result] Eisenkraft JB. Effects of anaesthetics on the pulmonary circulation. Br J Anaesth. 1990 Jul;65(1):63-78. doi: 10.1093/bja/65.1.63. No abstract available. PMID 2200486
- [Result] Lumb AB, Slinger P. Hypoxic pulmonary vasoconstriction: physiology and anesthetic implications. Anesthesiology. 2015 Apr;122(4):932-46. doi: 10.1097/ALN.0000000000000569. PMID 25587641
- [Result] Dunham-Snary KJ, Wu D, Sykes EA, Thakrar A, Parlow LRG, Mewburn JD, Parlow JL, Archer SL. Hypoxic Pulmonary Vasoconstriction: From Molecular Mechanisms to Medicine. Chest. 2017 Jan;151(1):181-192. doi: 10.1016/j.chest.2016.09.001. Epub 2016 Sep 16. PMID 27645688